CLINICAL TRIAL: NCT06535711
Title: Impact of Acute Computed Tomography on Treatment Decisions and Time to Intervention in Renal Colic
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-06913-01
Record Dates: First submitted 2024-07-23; First posted 2024-08-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute CT: Those with an acute CT (within 24 h).
  Interventions: Radiation: Acute CT
- Deferred CT: Those without an acute CT, instead a CT within 3-4 weeks.
  Interventions: Radiation: Deferred CT

INTERVENTIONS:
Radiation: Acute CT — Acute CT (a CT within 24 h)
  Groups: Acute CT
Radiation: Deferred CT — Deferred CT (a CT within 3-4 weeks)
  Groups: Deferred CT

SUMMARY:
This study intend to evaluate the use of acute computed tomography (CT) when acute renal colic, regarding treatment decisions, time to intervention and additional visits to the Emergency Department

DETAILED DESCRIPTION:
All patients with a diagnosis of urolithiasis at the Emergency Department in Helsingborg was included during one year, 1 July 2019 to 30 June 2020. Data regarding size and location of stone, treatment, follow up was extracted from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of urolithiasis at the Emergency Department in Helsingborg

Exclusion Criteria:

* Patients with a locked medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of urolithiasis at the Emergency Department during one year.
Sampling Method: Non-Probability Sample
Enrollment: 612 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Rate of interventions | 1 year
  Rate of ESWL (extracorporal shockwave lithotripsy), URS (ureteroscopy) and PCNL (percutanous nephrolithotripsy)
Time to intervention | 1 year
  Time to intervention, measured in number of days
Number of additional visits to the Emergency Department | 1 year
  Number of additional visits to the Emergency Department

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Wagenius, PhD, Principal Investigator — University of Lund, Sweden
Locations (1):
- Department of Urology, Helsingborg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Utter M, Altmark F, Popiolek M, Forsvall A, Lundstrom KJ, Thiel T, Wagenius M. Impact of emergency computed tomography on treatment and time to treatment for renal colic. Scand J Urol. 2025 Feb 5;60:29-35. doi: 10.2340/sju.v60.42593. PMID 39907293